CLINICAL TRIAL: NCT06036316
Title: Study of Language Disorders and Interactions Between Mnesic Capabilities and Semantic Competencies in Patients With Psychosis
Acronym: TDLRipsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Psychothérapique de Nancy (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-A00949-36
Record Dates: First submitted 2023-09-01; First posted 2023-09-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Psychosis; Schizophrenia; At-risk Mental State; Language Disorders
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Language Disorders | interventions — Psychiatric Status Rating Scales

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- early psychotic symptoms (Experimental): This group includes patients with ARMS and those with FEP. Although they are not in the same place in the continuum of psychosis, these patients benefit from the same language assessment and CAST, do not benefit from the TLC or the MINI, and the data from their neuropsychological and psychiatric assessment will be used , which is why we have chosen to bring them together in the same arm. They are between 16 and 35 years old and are cared for as part of their usual follow-up at the CPN (Nancy Psychotherapeutic Center). They must have received the diagnosis of ARMS and FEP according to the criteria of CAARMS and SPI-A.
  Interventions: Behavioral: Language assessment; Combination Product: CAST - Cannabis Abuse Screening Test
- patients with schizophrenia (Experimental): The schizophrenic patients group will benefit from language assessment, TLC and CAST. They are between 18 and 55 years old and are cared for as part of their usual follow-up at the CPN. They must have been diagnosed with schizophrenia according to DSM-5 (Diagnostic and Statistical Manual of Mental Disorders) criteria.
  Interventions: Behavioral: Language assessment; Behavioral: TLC - Scale for the Assessment of Thought, Language, and Communication; Combination Product: CAST - Cannabis Abuse Screening Test
- healthy controls (Experimental): The control group for this study will be made up of volunteers between the ages of 16 and 55, not suffering from any mental disorder detected on the MINI or from a developmental disorder of oral or written language. They will also benefit from an assessment of cannabis use using the CAST.
  Interventions: Behavioral: Language assessment; Behavioral: MINI - Mini International Neuropsychiatric Interview; Combination Product: CAST - Cannabis Abuse Screening Test

INTERVENTIONS:
Behavioral: Language assessment — The proposed speech and language therapy assessment will consist of a battery of standardized tests that speech and language therapists can use to assess the language skills in reception and expression of adult patients.
  Concerning the assessment of the interactions between working memory and semantic abilities, a complete protocol has been developed.
  Other Names: Speech and language therapy assessment
Behavioral: TLC - Scale for the Assessment of Thought, Language, and Communication — This scale is frequently used in psychiatry and is used to measure formal thought disorders in patients suffering from psychosis. As part of this study, it will be intended for patients suffering from schizophrenia
  Arms: patients with schizophrenia
Behavioral: MINI - Mini International Neuropsychiatric Interview — This scale corresponds to a rapid assessment of the psychiatric and psychological state of patients. It helps detect any psychiatric disorders. Here, it will be offered to volunteers who are part of the control group.
  Arms: healthy controls
Combination Product: CAST - Cannabis Abuse Screening Test — The purpose of this questionnaire is to approximate participants' cannabis consumption and to assess any disorders associated with cannabis consumption. It will be offered to all participants, patients and healthy controls

SUMMARY:
This research concerns the study of language disorders of patients present in the spectrum of psychosis. It is indeed accepted that psychotic disorders are associated with language difficulties, which are only poorly highlighted thanks to reusable tools in clinical practice. These language disorders impact communication, and concern many linguistic domains, thus covering phonology, lexicon, semantics, morphosyntax and pragmatics. It therefore seems relevant to characterize these language disorders and to assess to what extent they interact with the other symptoms of the pathology, in particular the course of the thought disorder and the neuropsychological symptoms. In addition, this study is particularly interested in the interactions between working memory capacities and those related to syntax. It is intended for different patients suffering from psychotic disorders of different intensities, treated in the Psychotherapeutic Center of Nancy. Patients suffering from at-risk mental state (ARMS), first episode of psychosis (FEP) or schizophrenia will benefit from a complete language assessment, evaluating each domain mentioned above, on the expressive and understanding sides. The results of the language assessment will be compared with those of a control group in the same tests. They will also be analyzed with regard to the neuropsychological and psychiatric elements noted in the patient's medical file, in order to highlight possible associations between language skills, neuropsychological and psychiatric symptoms in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* All Groups:

  * Patient affiliated or entitled to a social security scheme
  * Patient having received informed information on the study and having co-signed, with the investigator, a consent to participate in the study
  * For minor participants, at least one of the parents or holders of parental authority having been informed of the study, having received the information note relating to it and not having objected to the participation of his or her child
  * Native language: French
* ARMS and FEP Patient Group:

  * Age between 16 and 35 years old
  * Present the criteria for EMRP or FEP as defined by the Comprehensive Assessment of At Risk Mental State (CAARMS) or present the criteria for Disorders of the course of thought to the items of the Schizophrenia Proneness Instrument (SPI-A)
* Patients with schizophrenia group:

  * Age between 16 and 55 years old
  * Patient with diagnostic criteria for schizophrenia, as defined by DSM V (American Psychiatric Association, 2015)
  * Present the criteria for Disorganization of Speech and Formal Thought Disorder as defined by the Thinking, Language and Communication (TLC) Rating Scale.
* Healthy Volunteers Group:

  * Age between 16 and 55 years old
  * Parental authorization (of both parents) to participate in the study for minor patients

Exclusion Criteria:

* All groups:

  * Pregnant, parturient or nursing mother
  * Person deprived of liberty by a judicial or administrative decision
  * Person in a life-threatening emergency
  * Adult subject to a legal protection measure (guardianship, curatorship, safeguard of justice)
  * Adult person unable to express their consent and who is not the subject of a legal protection measure
  * Impairment of the subject making it difficult, if not impossible, for them to participate in the trial or to understand the information given to them
  * Abuse or dependence of any substance according to DSM V criteria excluding cannabis
* Healthy Volunteers Group:

  * Evolving psychiatric pathology (axis I of the DSM IV, measured at the MINI) excluding anxiety disorder
  * Presence of developmental disorder of oral language or written language revealed on clinical examination.

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2026-01-23 (Estimated); Study Completion 2026-01-23 (Estimated)

PRIMARY OUTCOMES:
language assessment performance score | day 1
  complete speech therapy assessment evaluating each language domain. and is based on the completion of a speech therapy assessment test and on the assessment of language abilities by the experimental speech therapist.

SECONDARY OUTCOMES:
CAARMS Speech Disorganization Severity Score | day 1
  CAARMS: Comprehensive Assessment of At Risk Mental State
Severity score for the disordered items of the course of thought of the SPI-A | day 1
  SPI-A:Schizophrenia Proneness Instrument
Severity score for speech disorganization and formal thought disorders on the TLC Scale | day 1
  TLC: Thinking, Language and Communication Rating Scale
Neuropsychological rating scales scores (CVLT) | day 1
  CVLT (California Verbal Learning test) (quantitative variable):
  CVLT: number of correct recognitions
Neuropsychological rating scales scores (CVLT total) | day 1
  CVLT (California Verbal Learning test) (quantitative variable):
  CVLT total: total number of words recalled during the test Recognition
Neuropsychological rating scales scores (Front and back spans) | day 1
  Front and back spans (quantitative variable) Front span size (number of digits recalled in front order)
Neuropsychological rating scales scores (Front and back spans 2) | day 1
  Front and back spans (quantitative variable) Reverse span size (number of digits recalled in reverse order)
Neuropsychological rating scales scores (TAP 1) | day 1
  TAP- Working Memory :Number of omissions TAP(Test of Attentional Performance) (quantitative variable)
Neuropsychological rating scales scores (TAP 2) | day 1
  TAP- Sustained attention :Number of omissions TAP(Test of Attentional Performance) (quantitative variable)
Neuropsychological rating scales scores (TAP 3) | day 1
  TAP- Flexibility :Number of errors TAP(Test of Attentional Performance) (quantitative variable)
Neuropsychological rating scales scores (TAP 4) | day 1
  TAP- Incompatibility TAP(Test of Attentional Performance) (quantitative variable)
Neuropsychological rating scales scores (TAP 5) | day 1
  TAP- Divided attention
Cannabis Abuse Screening Test (CAST) score | day 1
  CAST: Cannabis Abuse Screening Test

CONTACTS AND LOCATIONS:
Overall Officials: Florent Bernardin, PhD, Principal Investigator — Centre psychothérapeutique de Nancy
Locations (1):
- Centre Psychothérapeutique de Nancy, Laxou, France, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Majerus S. Language repetition and short-term memory: an integrative framework. Front Hum Neurosci. 2013 Jul 12;7:357. doi: 10.3389/fnhum.2013.00357. eCollection 2013. PMID 23874280